CLINICAL TRIAL: NCT00246285
Title: The Efficacy And Safety Of Risperidone In The Treatment Of Adolescents With Schizophrenia: A Six-Month Open-Label Study.
Brief Title: A Study of the Effectiveness and Safety of Risperidone in the Treatment of Adolescents With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR003364
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: schizophrenia; antipsychotic agents; risperidone; adolescents
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of the study is to assess the safety and effectiveness of risperidone (an antipsychotic medication) in adolescents with schizophrenia over 6 months of treatment.

DETAILED DESCRIPTION:
Although the safety and effectiveness of antipsychotic medications is well-established in adults with schizophrenia, these drugs have not been examined rigorously in adolescents with this disorder. Preliminary experience suggests that risperidone may hold promise for the treatment of these younger subjects. This is an open-label, multicenter trial of risperidone, formulated as an oral solution and tablets, in the treatment of adolescents with schizophrenia. It is an open-label, 6-month extension of two previous double-blind studies that assessed the safety and effectiveness of risperidone in the treatment of schizophrenia in an adolescent population. Patients may also enroll directly in this open-label trial. During the first week of the study, patients will receive increasing doses of risperidone to reach an optimal daily dose (2 to 6 mg/day), which will be maintained throughout the 6 months of the study. Assessments of effectiveness include the Positive and Negative Syndrome Scale for Schizophrenia (PANSS), a scale measuring the symptoms of schizophrenia, the Clinical Global Impression-Severity of Illness subscale (CGI-Severity), a scale measuring the severity of illness, the Clinical Global Impression-Improvement subscale (CGI-Improvement), a scale measuring clinical improvement, and the Children's Global Assessment Scale. Safety evaluations include the incidence of adverse events throughout the study, clinical laboratory tests (hematology, biochemistry, and urinalysis), vital signs (blood pressure, pulse, and temperature), weight, and electrocardiogram (ECG) recordings at specified intervals. The study hypothesis is that risperidone with be effective in the treatment of adolescents with schizophrenia, and well tolerated. Risperidone, oral solution (1 mg/ml) once daily; dose increasing from 0.01 mg/kg body weight (Day 1) to a range from 2 to 6 mg/day for 6 months. Oral tablets (0.5, 1, 2, 3, and 4 mg) once daily; dose increasing from 0.5 mg (Day 1) to a range of 2 to 6 mg/day for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia by criteria of Diagnostic and Statistical Manual of Mental Diseases, 4th edition (DSM-IV)
* expected to benefit from continuous treatment with risperidone, including patients who cannot tolerate their current antipsychotic therapy or are still exhibiting symptoms
* Positive and Negative Syndrome Scale for Schizophrenia (PANSS) score between 40 and 120 at start of study (not required for patients continuing from the 2 previous studies)

Exclusion Criteria:

* Meet criteria for other psychiatric disorders or mental retardation (documented IQ <70)
* history of substance dependence (including alcohol, but excluding nicotine and caffeine)
* hypersensitivity or intolerance to risperidone
* extrapyramidal symptoms (EPS) such as tremor that are not adequately controlled with medication

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 381 (Actual)
Dates: Start 2001-04; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change of Positive and Negative Syndrome Scale for Schizophrenia (PANSS) score from baseline to each visit during treatment; incidence of adverse events throughout study

SECONDARY OUTCOMES:
Clinical Global Impression-Severity of Illness (CGI-Severity) and Clinical Global Impression-Improvement (CGI-Improvement) at each visit; Children's Global Assessment Scale at start and end of study; clinical laboratory tests, vital signs, weight, ECGs.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Pandina G, Kushner S, Karcher K, Haas M. An open-label, multicenter evaluation of the long-term safety and efficacy of risperidone in adolescents with schizophrenia. Child Adolesc Psychiatry Ment Health. 2012 Jun 7;6(1):23. doi: 10.1186/1753-2000-6-23. PMID 22676070
- See also: A Study of the Effectiveness and Safety of Risperidone in the Treatment of Adolescents With Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=522&filename=CR003364_CSR.pdf